CLINICAL TRIAL: NCT04547426
Title: Metabolic Effects of Snuff and Red Wine
Brief Title: Effects of Snuff and/or Red Wine om Metabolic Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, professor, MD, University Hospital, Linkoeping
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EPN2020-00839
Record Dates: First submitted 2020-08-31; First posted 2020-09-14 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Metabolic Rate; Hunger; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Wine; Ethanol; Tobacco, Smokeless; Nicotine

STUDY DESIGN:
Who Masked: Participant
Masking Description: We use non-alcoholic or alcohol containing wine and regular or nicotine free snuff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- red wine and snuff (Active Comparator): regular red wine and moist snuff
  Interventions: Other: Wine with or without alcohol and snuff with or without nicotine
- red wine and nicotine-free snuff (Active Comparator): regular red wine and nicotine-free snuff
  Interventions: Other: Wine with or without alcohol and snuff with or without nicotine
- non alcoholic red wine and regular moist snuff (Active Comparator): non alcoholic red wine and regular moist snuff with nicotine
  Interventions: Other: Wine with or without alcohol and snuff with or without nicotine
- non-alcoholic red wine and nicotine-free snuff (Placebo Comparator): Non-alcoholic red wine and nicotine-free snuff
  Interventions: Other: Wine with or without alcohol and snuff with or without nicotine

INTERVENTIONS:
Other: Wine with or without alcohol and snuff with or without nicotine — Two by two factorial of wine and snuff with meals

SUMMARY:
About 14 healthy participants, consume a standardized breakfast combined with either using regular or nicotine-free moist snuff. The metabolic rate is measured every hour for four hours on each occasion starting in the morning. Participants are also randomized to get red wine or non-alcoholic red wine to the meal.

DETAILED DESCRIPTION:
About 14 healthy participants, consume a standardized breakfast combined with either using regular or nicotine-free moist snuff. The metabolic rate is measured measured before the meal and then every hour for a total of four hours on each occasion that starts in the morning. Participants are also randomized to get red wine or non-alcoholic red wine to the meal. Since there are four possible combinations of the wine and the snuff, all participants do the test on four occasions. Except for metabolic rate we will also analyze hormone responses regarding appetite or hunger.

ELIGIBILITY:
Inclusion Criteria: No significant disease -

Exclusion Criteria: known illnesses, thyroid disease, need to take prednisolone, psychiatric disease,inability to understand Swedish

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
level of metabolic rate | 4 hours
  Measurement of metabolic rate by registration of CO2 in breath and the oxygen uptake

SECONDARY OUTCOMES:
sense of appetite | 4 hours
  determination of the hormones ghrelin and GLP-1 in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine and Health Sciences, Linköping, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No
There are no such plans